CLINICAL TRIAL: NCT04305756
Title: Impact of Prophylactic Low-molecular Weight Heparin Dosing on Clotting Parameters Following Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Torri Metz, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 130494
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Thromboembolism; Postpartum DVT; Thrombosis
Keywords: Factor Xa; Biomarkers; Enoxaparin
MeSH Terms: conditions — Thromboembolism; Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight-based LMWH (Experimental): Participants will receive a weight-based dose of prophylactic enoxaparin.
  - For all BMI groups: 0.5mg/kg rounded to the nearest 10mg will be injected subcutaneously every 12 hours
  Interventions: Drug: Enoxaparin
- Fixed LMWH (Active Comparator): Participants will receive a fixed dose of prophylactic enoxaparin.
  * For BMI <40: 40mg injected subcutaneously every 24 hours
  * For BMI > or = to 40: 40mg injected subcutaneously every 12 hours
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Low molecular weight heparin
  Other Names: Lovenox

SUMMARY:
The aim of this study is to evaluate the efficacy of two dosing regimens of low molecular weight heparin (LMWH) to reach prophylactic anti-factor Xa levels in post-cesarean delivery women. Half of participants will receive a fixed dose of LMWH, while the other half will receive a weight-based dose. The hypothesis is that the use of a weight-based dose will result in more women reaching prophylactic levels.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a major contributor to maternal morbidity and mortality. The immediate postpartum period is a high risk time for VTE, and cesarean delivery is an additional risk factor. In the United States, use of postpartum VTE prophylaxis with low-molecular weight heparin (LMWH) is commonly used but without a standard protocol or dose across all hospitals. A fixed-dose of LMWH is frequently used based on data from non-obstetric studies. However, there are concerns that in the postpartum population this fixed dose may not be adequate for prophylaxis.

This study aims to evaluate the efficacy of fixed dose versus weight-based LMWH to reach prophylactic anti-Xa levels in post-cesarean delivery women. This will be a randomized controlled trial (RCT) with half of participants receiving a fixed dose of LMWH and half of participants receiving a weight-based dose of LMWH. The hypothesis is that the use of a weight-based LMWH compared to a fixed dose will result in more women achieving prophylactic anti-Xa levels.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery
* Meet facility guidelines for postpartum venous thromboembolism (VTE) prophylaxis: Presence of 1 major, or 2 or more moderate, risk factors.
* Major risk factors: history of venous thromboembolism, high risk thrombophilia, BMI ≥40, high risk medical comorbidities (heart disease, sickle cell disease, systemic lupus erythematosus, inflammatory bowel disease), cesarean hysterectomy, nephrotic range proteinuria, or cesarean intrapartum/during labor
* Moderate risk factors: BMI > 30, multifetal pregnancy, postpartum hemorrhage (>1L blood loss), tobacco use, non-laboring or elective cesarean, preeclampsia, infection, preterm delivery (< 37 weeks gestational age), age > 35 years, low risk thrombophilia, family history of venous thromboembolism, stillbirth, varicose veins, prolonged labor (> 24 hours)

Exclusion Criteria:

* Contraindication to anticoagulation
* Plan for therapeutic anticoagulation (antepartum or postpartum)
* Known renal dysfunction (Creatinine clearance < 30 mL/minute)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Prophylactic peak anti-Xa level | Postoperative day #3 at peak (4-6 hours post-dose)
  Anti-Xa level in prophylactic range (0.2 to 0.6 IU/mL)

SECONDARY OUTCOMES:
Venous thromboembolism | From delivery through 6 weeks postpartum
  Presence of venous thromboembolism as confirmed on diagnostic imaging
Wound Complications | From delivery through 6 weeks postpartum
  Post-cesarean wound hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Torri Metz, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Bruno AM, Allshouse AA, Campbell HM, Branch DW, Lim MY, Silver RM, Metz TD. Weight-Based Compared With Fixed-Dose Enoxaparin Prophylaxis After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2022 Oct 1;140(4):575-583. doi: 10.1097/AOG.0000000000004937. Epub 2022 Sep 7. PMID 36075079